CLINICAL TRIAL: NCT06262490
Title: Impact of Pelvic Floor Rehabilitation Combined With Ultrasound Therapy on Osteomyoarticular Symptoms in Chronic Perineal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya T- Allah Mohamed Nabil Mohamed, PhD student at Department of Physical Therapy for Women's Health, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004765
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Chronic Perineal Pain; Pelvic Floor Disorders
Keywords: Pelvic floor rehabilitation; Ultrasound; Osteomyoarticular symptoms; Chronic Perineal pain
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group A (Active Comparator): They will receive traditional ultrasound therapy for six weeks
  Interventions: Device: Traditional ultrasound therapy
- Study group B (Experimental): They will receive the same traditional ultrasound therapy in addition to pelvic floor rehabilitation for six weeks
  Interventions: Device: Traditional ultrasound therapy; Other: Pelvic floor rehabilitation

INTERVENTIONS:
Device: Traditional ultrasound therapy — Ultrasound therapy for 2 session per week for until completing 12 treatment sessions (six weeks) with frequencies up to 3 MHz are used clinically to promote healing
Other: Pelvic floor rehabilitation — Pelvic floor rehabilitation for 3 sessions per week for (six weeks) until completing 18 sessions with sessions lasting between 30-45 minutes
  Arms: Study group B

SUMMARY:
The purpose of the study is to find out the effect of pelvic floor rehab combined with ultrasound have effect in chronic perineal pain subjects associated with osteomyoarticular symptoms .

DETAILED DESCRIPTION:
Chronic perineal pain is the anorectal and perineal pain without underlying organic disease, anorectal or endopelvic, which has been excluded by careful physical examination, radiological and endoscopic investigations. So, perineal and vaginal pain after vaginal delivery has been associated with tissue trauma related to operative vaginal delivery, perineal laceration, and episiotomy.

Studies assessing chronic pain after vaginal delivery report 2% to 10% of women with pain at six months and later, almost exclusively in mothers who had an assisted vaginal birth. Postpartum pain intensity is usually higher when it is related to vaginal delivery than to cesarean delivery and more severely affects the woman's quality of life and mood.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subjects will be ranged from 20 to 35 years.
2. All participants had vaginal delivery with episiotomy.
3. They are in late post partum period over 6 months
4. Their BMI will be ranger from 25 to 30 kg/m2.
5. All participants have mechanical low back pain.
6. All participants have perineal pain.
7. The Number of parity Ranged from 2-3 times.

Exclusion Criteria:

1. Females will be excluded if they have any spine or lower extremities injuries or previous surgeries.
2. Females with radicular back pain.
3. Inability to understand the written and verbal instruction.
4. Females had irregular menstrual cycle

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of osteomyoarticular symptoms | 6 weeks
  It will be assessed before and after the end of treatment for each participant in both groups using Nordic Musculoskeletal Questionnaire (NMQ), an instrument characterized by multiple or binary choices facing osteomyoarticular symptoms in various anatomical regions that these symptoms appear more frequently, and a questionnaire that has good reliability (Legault et al., 2014).
Assessment of perineal pain intensity | 6 weeks
  It will be assessed before and after the end of treatment for each participant in both groups through the visual analouge scale (VAS). It is a 10-cm horizontal line on which the patient's pain intensity was represented by a point between the extremes of "no pain at all" and "worst pain imaginable". Its simplicity, reliability and validity, as well as its ratio scale properties, make the VAS the optimal tool for describing pain intensity. Each participant will be asked to mark a point on the VAS line between the extremes that related to her perineal intensity. Then, the centimeters will be measured in each time from the left end of the line to the marked point to obtain the VAS score for perineal pain intensity

SECONDARY OUTCOMES:
Assessment of pelvic floor muscle strength | 6 weeks
  It will be assessed before and after the end of treatment for each participant in both groups by Kegel perineometer
Assessment of pelvic floor muscle tightness | 6 weeks
  It will be assessed before and after the end of treatment for each participant in both groups by the manual pelvic floor muscle examination
Assessment of lumbar spine mobility | 6 weeks
  It will be assessed before and after the end of treatment for each participant in both groups by the modified Schober test

CONTACTS AND LOCATIONS:
Overall Officials: Salwa M. El Badry, Prof., Study Chair — Department of Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.; Amel M. Yousef, Study Director — Department of Physical Therapy for Woman's Health, Faculty of physical therapy, Cairo University, Giza, Egypt.
Locations (1):
- Cairo University, Giza, Egypt